CLINICAL TRIAL: NCT05903924
Title: Motion Serifos: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy of Tradipitant in Participants Affected by Motion Sickness During Travel
Brief Title: Motion Serifos: A Study to Investigate the Efficacy of Tradipitant in Participants Affected by Motion Sickness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VLY-686-3404
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Results first posted 2025-04-04 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Tradipitant High Dose (Experimental)
  Interventions: Drug: Tradipitant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Tradipitant Low Dose (Experimental)
  Interventions: Drug: Tradipitant

INTERVENTIONS:
Drug: Tradipitant — Oral Capsule
  Arms: Tradipitant High Dose; Tradipitant Low Dose
Drug: Placebo — Oral Capsule
  Arms: Placebo

SUMMARY:
A multi-center, randomized, double-blind, placebo-controlled study to investigate the efficacy of tradipitant in participants affected by motion sickness during travel

ELIGIBILITY:
Inclusion Criteria:

* History of motion sickness
* Age 18-75

Exclusion Criteria:

* Nausea-inducing disorder other than motion sickness
* BMI>40
* History of intolerance and/or hypersensitivity to Neurokinin-1 Receptor antagonists

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2023-09-09 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-04-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Pacific Research Partners, San Diego, California
  - Lumos Clinical Research, San Jose, California
  - Santa Monica Clinical Trials, Santa Monica, California
  - Beacon Clinical Research, Boston, Massachusetts
  - Manhattan Medical Research, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tradipitant High Dose | Tradipitant Low Dose | Placebo
Started | 106 | 104 | 106
Completed | 105 | 104 | 106
Not Completed | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tradipitant High Dose | Tradipitant Low Dose | Placebo | Total
Number analyzed (Participants) | 106 | 104 | 106 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (14.67) | 47.3 (14.31) | 45.3 (14.86) | 46.3 (14.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 62 | 60 | 178
  Male | 50 | 42 | 46 | 138
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 16 | 16 | 43
  Not Hispanic or Latino | 91 | 84 | 82 | 257
  Unknown or Not Reported | 4 | 4 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaskan Native | 0 | 0 | 1 | 1
  Race: Asian | 15 | 9 | 12 | 36
  Race: Black or African American | 5 | 4 | 6 | 15
  Race: Native Hawaiian or Pacific Islander | 2 | 0 | 0 | 2
  Race: White | 80 | 88 | 78 | 246
  Race: Other | 1 | 1 | 5 | 7
  Race: Multiple | 3 | 2 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 106 | 104 | 106 | 316
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.453 (5.0221) | 26.989 (4.0170) | 26.811 (4.3017) | 27.085 (4.4638)

OUTCOME MEASURES:

1. Primary Outcome: Prevention of Vomiting Measured by Vomiting Assessment (VA)
Description: Prevention of vomiting measured by Vomiting Assessment (VA) score. The VA is a 1-item questionnaire to objectively measure the incidence of emesis. Participants will indicate whether or not they have vomited.
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Tradipitant High Dose | Tradipitant Low Dose | Placebo
Number analyzed (Participants) | 106 | 104 | 106
Participants | 11 | 19 | 40

ADVERSE EVENTS:
Time Frame: Adverse Events were recorded from time of randomization until the end of study visit, up to 7 days.
Arm/Group | Tradipitant High Dose | Tradipitant Low Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/106 | 0/104 | 0/106
Serious Adverse Events (participants affected / at risk) | 0/106 | 0/104 | 0/106
Other Adverse Events (participants affected / at risk) | 29/106 | 24/104 | 19/106
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tradipitant High Dose (N=106) | Tradipitant Low Dose (N=104) | Placebo (N=106)
Headache (Nervous system disorders) | 10 | 9 | 9
Somnolence (Nervous system disorders) | 9 | 6 | 8
Fatigue (General disorders) | 12 | 9 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT05903924/Prot_SAP_000.pdf